CLINICAL TRIAL: NCT02329171
Title: TOPical Imiquimod Treatment of High-grade Cervical Intraepithelial Neoplasm: a Randomized Controlled Trial.
Brief Title: Imiquimod Treatment of CIN Lesions
Acronym: TOPIC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient number of participants.
Sponsor: Maastricht University Medical Center (Other)
Collaborators: MEDA Pharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METC 13-2-031
Record Dates: First submitted 2014-12-22; First posted 2014-12-31 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2016-06

CONDITIONS: Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Imiquimod treatment arm (Experimental): Patients in this group will be treated with imiquimod during 16 weeks. Colposcopy with diagnostic biopsies will be performed after 10 weeks. In case of progressive disease, the treatment will be ended and appropriate surgical excision will be performed. Treatment efficacy will be evaluated after 20 weeks, by colposcopy with diagnostic biopsies.
  Interventions: Drug: Imiquimod
- Standard treatment arm (Active Comparator): Large loop excision of the transformation zone (LLETZ) will be performed in this group, as standard treatment.
  Interventions: Procedure: LLETZ

INTERVENTIONS:
Drug: Imiquimod — Imiquimod 5% cream will be administered in a vaginal applicator, containing 12,5 mg of imiquimod (one sachet). The cream will be self-administered three times per week, by use of a vaginal applicator.
  Other Names: Imiquimod, Aldara.
  Arms: Imiquimod treatment arm
Procedure: LLETZ — Standard treatment consists of a LLETZ procedure, in which excision of the transformation zone and macroscopic lesions is performed by a monopolar loop electrode, under local anaesthesia. The excision is usually performed in two or three steps, depending on the size of the lesions.
  Other Names: Loop excision
  Arms: Standard treatment arm

SUMMARY:
Rationale:

Cervical Intraepithelial Neoplasia (CIN) is the premalignant condition of cervical cancer. High grade CIN (CIN 2-3) is currently treated by large loop excision of the transformation zone (LLETZ). This treatment has potential complications, such as hemorrhage, infection and preterm birth in subsequent pregnancies. For this reason, non-invasive therapies are needed. Imiquimod (an immunomodulator) was proven effective in the treatment of HPV-related vulvar intraepithelial neoplasia (VIN) and may also be effective in HPV-related CIN. [van Seters, 2012] However, the evidence is limited and study results are not consistent. [Grimm, 2012; Pachman, 2012; Lin, 2012]

Objectives:

Primary objectives: (1) to investigate the efficacy of imiquimod 5% cream for the treatment of CIN2-3 lesions and (2) to develop biomarker panels to predict clinical response to imiquimod therapy.

Secondary objectives: to assess side effects of imiquimod treatment and LLETZ, disease recurrence and quality of life.

Hypothesis:

The investigators hypothesize that imiquimod will be an effective treatment modality in approximately 50-75% of CIN lesions treated without surgical intervention.

Study design:

Single-centre randomized controlled intervention trial.

Study population:

140 women with a histological diagnosis of CIN2-3, equally divided over two study arms.

Intervention:

Patients will be randomized into one of two arms:

1. Imiquimod treatment arm. Patients in this group are treated by a 16-week regime of imiquimod 5% cream.
2. Standard treatment arm. LLETZ will be performed on patients in this group.

Colposcopy with diagnostic biopsies will be performed after 10 weeks for the imiquimod treatment arm. In case progressive disease, the treatment will be ended and appropriate surgical excision will be performed. Treatment efficacy will be evaluated after 20 weeks, by colposcopy with diagnostic biopsies. A histological biomarker panel will be developed, consisting of markers representing both host and viral factors.

Main study parameters/endpoints:

The primary endpoint of the study is regression-or-not of CIN2-3, defined as CIN1 or less at the colposcopy at 20 weeks for the imiquimod arm and PAP 1 cytology at 6 months for the LLETZ group.

DETAILED DESCRIPTION:
The treatment period was set at 20 weeks, in order to realize adequate treatment efficacy of imiquimod, while minimizing the risk of progression of cervical dysplasia to invasive disease in the conservative treatment group. Based on the available literature on the natural history of CIN and several studies on cervical dysplasia that included a conservative treatment group, the risk of disease progression within the treatment period of 20 weeks is estimated to be marginal. Approximately 30% of high-grade CIN progresses to cervical cancer. [Peto, 2004; McCredie, 2008]. This is believed to be a slow process, which can take many years. The annual risk of progression of CIN 3 to invasive cervical cancer is estimated to be less than 1%.[Canfell, 2004]. Ten studies were identified in which a total of 637 patients with high grade CIN were included either as a control group, receiving conservative treatment during 6 weeks to 15 months, or followed during the period between diagnosis and LLETZ.[Grimm, 2012, Follen, 2001; Meyskens, 1994; Keefe, 2001; Alvarez, 2003; Garcia, 2004; Van Pachterbeke, 2009; Kaufmann, 2007; Trimble 2005; Munk, 2012] Three cases of invasive disease were identified: all occured in the same study after 16 weeks of conservative treatment. Other studies showed no progression to invasive disease. One case of progression was reported with undefined disease grade and follow-up term. The possibility of invasive disease already present at the initial colposcopy (biopsy error) cannot be excluded. Based on these results, the investigators selected a treatment period of 20 weeks, with a control colposcopy with diagnostic biopsies after ten weeks.

The current study protocol includes a substantial amendment to the original study protocol, which consisted of three study arms: imiquimod treatment arm, LLETZ treatment arm and an observational arm. The purpose of the observational arm was to assess spontaneous regression of high-grade CIN and to develop a prognostic biomarker panel to predict spontaneous regression of high-grade CIN. Patients in the observational arm underwent no treatment for a period of maximum 20 weeks. Histological assessment of disease development was performed after 10 and 20 weeks by colposcopy with diagnostic biopsies. Inclusion of patients into the study was hampered by the observational arm: patients declined the study because they wished to be treated, rather than undergo observational management. The observational arm was removed from the study.

ELIGIBILITY:
Inclusion criteria:

* newly diagnosed high grade CIN lesions (CIN 2-3), histologically confirmed
* age 18 years or older

Exclusion criteria:

* immunodeficiency
* pregnancy or lactation
* legally incapability
* history of histologically conformed high-grade CIN

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy: histological disease regression | 20 weeks
  Defined as following:
  * for imiquimod treatment arm: CIN1 or less in diagnostic biopsies at colposcopy at 20 weeks
  * for LLETZ arm: PAP 1 at 6 months follow-up
Baseline biomarker profile predicting clinical response to imiquimod treatment | 20 weeks
  The biomarker profiles will consist of markers reflecting host and viral factors, including HPV-genotype, markers of immunologic response (CD4, CD8, CD25, CD138, Fox p3) and markers of cell cycle processes (Rb, p53, Ki67, CK 13/14, IMP3).

SECONDARY OUTCOMES:
Prevalence and severity of side effects of imiquimod and LLETZ treatment | 6 weeks, 10 weeks, 14 weeks and 20 weeks for imiquimod treatment and 6 weeks for LLETZ treatment
  The prevalence and severity of side effects of imiquimod and LLETZ treatment, as documented according to Common Terminology Criteria for Adverse Events guidelines.
Quality of life for all treatment groups. | Baseline, 20 weeks and 1 year
  Assessed by the following questionnaires: RAND 36, EORTC QLQ-C30 and EORTC QLQ-CX24.
Disease recurrence for all treatment groups. | 6, 12 and 24 months
  Defined as abnormal cervical cytology.

CONTACTS AND LOCATIONS:
Overall Officials: Arnold J Kruse, MD, PhD, Study Director — Maastricht University Medical Center; R.F.P.M. Kruitwagen, Professor, Study Chair — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

REFERENCES:
- [Background] van Seters M, van Beurden M, ten Kate FJ, Beckmann I, Ewing PC, Eijkemans MJ, Kagie MJ, Meijer CJ, Aaronson NK, Kleinjan A, Heijmans-Antonissen C, Zijlstra FJ, Burger MP, Helmerhorst TJ. Treatment of vulvar intraepithelial neoplasia with topical imiquimod. N Engl J Med. 2008 Apr 3;358(14):1465-73. doi: 10.1056/NEJMoa072685. PMID 18385498
- [Background] Grimm C, Polterauer S, Natter C, Rahhal J, Hefler L, Tempfer CB, Heinze G, Stary G, Reinthaller A, Speiser P. Treatment of cervical intraepithelial neoplasia with topical imiquimod: a randomized controlled trial. Obstet Gynecol. 2012 Jul;120(1):152-9. doi: 10.1097/AOG.0b013e31825bc6e8. PMID 22914404
- [Background] Pachman DR, Barton DL, Clayton AC, McGovern RM, Jefferies JA, Novotny PJ, Sloan JA, Loprinzi CL, Gostout BS. Randomized clinical trial of imiquimod: an adjunct to treating cervical dysplasia. Am J Obstet Gynecol. 2012 Jan;206(1):42.e1-7. doi: 10.1016/j.ajog.2011.06.105. Epub 2011 Jul 13. PMID 21907959
- [Background] Lin CT, Qiu JT, Wang CJ, Chang SD, Tang YH, Wu PJ, Jung SM, Huang CC, Chou HH, Jao MS, Lai CH. Topical imiquimod treatment for human papillomavirus infection in patients with and without cervical/vaginal intraepithelial neoplasia. Taiwan J Obstet Gynecol. 2012 Dec;51(4):533-8. doi: 10.1016/j.tjog.2012.09.006. PMID 23276555
- [Background] Peto J, Gilham C, Deacon J, Taylor C, Evans C, Binns W, Haywood M, Elanko N, Coleman D, Yule R, Desai M. Cervical HPV infection and neoplasia in a large population-based prospective study: the Manchester cohort. Br J Cancer. 2004 Aug 31;91(5):942-53. doi: 10.1038/sj.bjc.6602049. PMID 15292939
- [Background] McCredie MR, Sharples KJ, Paul C, Baranyai J, Medley G, Jones RW, Skegg DC. Natural history of cervical neoplasia and risk of invasive cancer in women with cervical intraepithelial neoplasia 3: a retrospective cohort study. Lancet Oncol. 2008 May;9(5):425-34. doi: 10.1016/S1470-2045(08)70103-7. Epub 2008 Apr 11. PMID 18407790
- [Background] Canfell K, Barnabas R, Patnick J, Beral V. The predicted effect of changes in cervical screening practice in the UK: results from a modelling study. Br J Cancer. 2004 Aug 2;91(3):530-6. doi: 10.1038/sj.bjc.6602002. PMID 15266332
- [Background] Follen M, Atkinson EN, Schottenfeld D, Malpica A, West L, Lippman S, Zou C, Hittelman WN, Lotan R, Hong WK. A randomized clinical trial of 4-hydroxyphenylretinamide for high-grade squamous intraepithelial lesions of the cervix. Clin Cancer Res. 2001 Nov;7(11):3356-65. PMID 11705848
- [Background] Meyskens FL Jr, Surwit E, Moon TE, Childers JM, Davis JR, Dorr RT, Johnson CS, Alberts DS. Enhancement of regression of cervical intraepithelial neoplasia II (moderate dysplasia) with topically applied all-trans-retinoic acid: a randomized trial. J Natl Cancer Inst. 1994 Apr 6;86(7):539-43. doi: 10.1093/jnci/86.7.539. PMID 8133537
- [Background] Keefe KA, Schell MJ, Brewer C, McHale M, Brewster W, Chapman JA, Rose GS, McMeeken DS, Lagerberg W, Peng YM, Wilczynski SP, Anton-Culver H, Meyskens FL, Berman ML. A randomized, double blind, Phase III trial using oral beta-carotene supplementation for women with high-grade cervical intraepithelial neoplasia. Cancer Epidemiol Biomarkers Prev. 2001 Oct;10(10):1029-35. PMID 11588128
- [Background] Alvarez RD, Conner MG, Weiss H, Klug PM, Niwas S, Manne U, Bacus J, Kagan V, Sexton KC, Grubbs CJ, Eltoum IE, Grizzle WE. The efficacy of 9-cis-retinoic acid (aliretinoin) as a chemopreventive agent for cervical dysplasia: results of a randomized double-blind clinical trial. Cancer Epidemiol Biomarkers Prev. 2003 Feb;12(2):114-9. PMID 12582020
- [Background] Garcia F, Petry KU, Muderspach L, Gold MA, Braly P, Crum CP, Magill M, Silverman M, Urban RG, Hedley ML, Beach KJ. ZYC101a for treatment of high-grade cervical intraepithelial neoplasia: a randomized controlled trial. Obstet Gynecol. 2004 Feb;103(2):317-26. doi: 10.1097/01.AOG.0000110246.93627.17. PMID 14754702
- [Background] Van Pachterbeke C, Bucella D, Rozenberg S, Manigart Y, Gilles C, Larsimont D, Vanden Houte K, Reynders M, Snoeck R, Bossens M. Topical treatment of CIN 2+ by cidofovir: results of a phase II, double-blind, prospective, placebo-controlled study. Gynecol Oncol. 2009 Oct;115(1):69-74. doi: 10.1016/j.ygyno.2009.06.042. Epub 2009 Aug 3. PMID 19647859
- [Background] Kaufmann AM, Nieland JD, Jochmus I, Baur S, Friese K, Gabelsberger J, Gieseking F, Gissmann L, Glasschroder B, Grubert T, Hillemanns P, Hopfl R, Ikenberg H, Schwarz J, Karrasch M, Knoll A, Kuppers V, Lechmann M, Lelle RJ, Meissner H, Muller RT, Pawlita M, Petry KU, Pilch H, Walek E, Schneider A. Vaccination trial with HPV16 L1E7 chimeric virus-like particles in women suffering from high grade cervical intraepithelial neoplasia (CIN 2/3). Int J Cancer. 2007 Dec 15;121(12):2794-800. doi: 10.1002/ijc.23022. PMID 17721997
- [Background] Trimble CL, Piantadosi S, Gravitt P, Ronnett B, Pizer E, Elko A, Wilgus B, Yutzy W, Daniel R, Shah K, Peng S, Hung C, Roden R, Wu TC, Pardoll D. Spontaneous regression of high-grade cervical dysplasia: effects of human papillomavirus type and HLA phenotype. Clin Cancer Res. 2005 Jul 1;11(13):4717-23. doi: 10.1158/1078-0432.CCR-04-2599. PMID 16000566
- [Background] Munk AC, Gudlaugsson E, Ovestad IT, Lovslett K, Fiane B, Hidle Bv, Kruse AJ, Skaland I, Janssen EA, Baak JP. Interaction of epithelial biomarkers, local immune response and condom use in cervical intraepithelial neoplasia 2-3 regression. Gynecol Oncol. 2012 Dec;127(3):489-94. doi: 10.1016/j.ygyno.2012.09.010. Epub 2012 Sep 24. PMID 23017821
- [Derived] Koeneman MM, Kruse AJ, Kooreman LF, Zur Hausen A, Hopman AH, Sep SJ, Van Gorp T, Slangen BF, van Beekhuizen HJ, van de Sande AJ, Gerestein CG, Nijman HW, Kruitwagen RF. Preliminary stop of the TOPical Imiquimod treatment of high-grade Cervical intraepithelial neoplasia (TOPIC) trial. BMC Cancer. 2017 Feb 7;17(1):110. doi: 10.1186/s12885-017-3108-9. PMID 28173776
- [Derived] Koeneman MM, Kruse AJ, Kooreman LFS, Zur Hausen A, Hopman AHN, Sep SJS, Van Gorp T, Slangen BFM, van Beekhuizen HJ, van de Sande M, Gerestein CG, Nijman HW, Kruitwagen RFPM. TOPical Imiquimod treatment of high-grade Cervical intraepithelial neoplasia (TOPIC trial): study protocol for a randomized controlled trial. BMC Cancer. 2016 Feb 20;16:132. doi: 10.1186/s12885-016-2187-3. PMID 26897518